CLINICAL TRIAL: NCT02667262
Title: An Observational Study to Develop Computable Algorithms for Identifying Opioid Abuse and Addiction Based on Administrative Claims Data
Brief Title: An Observational Study to Develop Algorithms for Identifying Opioid Abuse and Addiction Based on Admin Claims Data
Status: Completed | Type: Observational
Sponsor: Member Companies of the Opioid PMR Consortium (Industry)
Collaborators: World Health Information Science Consultants, LLC (Other); Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: Observational Study 3033-7; 3033-7 (Other: Member Companies of the Opioid PMR Consortium)
Record Dates: First submitted 2016-01-18; First posted 2016-01-28 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Opioid-Related Disorders; Opiate Addiction; Narcotic Abuse; Drug Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Extended Release and/or Long-Acting Opioids
  Interventions: Other: Algorithm to identify patients experiencing opioid abuse/addiction

INTERVENTIONS:
Other: Algorithm to identify patients experiencing opioid abuse/addiction

SUMMARY:
The purpose of this study is to develop and validate a classification model based entirely on medical claims data that can be used to identify patients experiencing prescription opioid abuse/addiction among patients receiving extended-release (ER) and/or long-acting (LA) opioids

DETAILED DESCRIPTION:
The most widely available information about patient care and conditions is that contained in medical claims data. If such data can be used to develop a model for identifying patients experiencing prescription opioid abuse/addiction it could be widely applied to patient populations throughout the United States.

A study recently conducted at Group Health comparing International Classification of Disease, Ninth edition (ICD-9) coding for opioid abuse/addiction to textual mentions in clinical notes describing abuse/addiction found that ICD-9 codes were 64% sensitive and 96% specific in their ability to identify patients experiencing opioid abuse/addiction (compared to evidence from clinical notes). This Group Health study considered codes for abuse (305.x) and addiction (304.x) equivalent because clinicians' usage of these codes did not differentiate well between abuse and addiction.

Needed are methods that can accurately identify patients experiencing opioid abuse/addiction based on widely available claims data.

This study will not evaluate opioid misuse because this will be captured by instruments in a prospective study of pain patients (Study 1A) using a combination of adapted validated instruments, and other new instruments that will be evaluated in post-marketing requirement (PMR) Study 2, plus medical record review to supplement questionnaire-based measurement of misuse, abuse and addiction with aberrant behaviors and physician text entries in the medical records.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Receipt of at least a 60 day's supply of ER/LA opioid analgesics within a 90-day period (including transdermal or oral opioids but excluding buprenorpine)
3. Minimum of at least two years continuous enrollment in Group Health integrated group practice (IGP)

Exclusion Criteria:

1. Residence in a nursing home at any time during the study period
2. Enrollment in a hospice care program at any time during the study period

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with at least two years continuous enrollment in Group Health integrated group practice (IGP) receiving ER/LA opioid analgesics
Sampling Method: Probability Sample
Enrollment: 1667 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Opioid abuse/addiction | Retrospective review of data from 2006 to 2015, up to 9 years
  This will be assessed from three data sources: a diagnostic algorithm that uses coded terms in claims data, Natural Language Processing assessment of text in electronic medical records, and medical chart review by clinicians trained in chart review

CONTACTS AND LOCATIONS:
Overall Officials: Paul Coplan, MS, ScD, MBA, Study Chair — Purdue Pharma LP

REFERENCES:
- [Derived] Carrell DS, Albertson-Junkans L, Ramaprasan A, Scull G, Mackwood M, Johnson E, Cronkite DJ, Baer A, Hansen K, Green CA, Hazlehurst BL, Janoff SL, Coplan PM, DeVeaugh-Geiss A, Grijalva CG, Liang C, Enger CL, Lange J, Shortreed SM, Von Korff M. Measuring problem prescription opioid use among patients receiving long-term opioid analgesic treatment: development and evaluation of an algorithm for use in EHR and claims data. J Drug Assess. 2020 Apr 28;9(1):97-105. doi: 10.1080/21556660.2020.1750419. eCollection 2020. PMID 32489718